CLINICAL TRIAL: NCT05707858
Title: The Naples Pediatric Food Allergy (NAPFA) Score
Acronym: NAPFA
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Professor of Pediatrics, Federico II University
Other Study IDs: 284/21
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Food Allergy in Children
Keywords: Food allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject with suspected food allergy
  Interventions: Other: Development of the NAPFA score

INTERVENTIONS:
Other: Development of the NAPFA score — In subjects with suspected food allergy we will evaluate main anamnestic, and clinical features to develop the NAPFA score

SUMMARY:
Food Allergy (FA) is one of the most expensive allergic disorders in the pediatric age, and affecting up to 10% of children worldwide, it is recognized as a global health problem. The Oral Food Challenge (OFC) is the gold standard for FA diagnosis, but it is time-consuming, expensive, and potentially dangerous, as it can determine severe anaphylaxis. In addition, causing long-lasting impact on patient anxiety and mental health due to the physical duress and health risks involved with its application, OFC strategy is little applied in clinical practice with consequent diagnostic errors and delays. The goal of the Naples Pediatric Food Allergy (NAPFA) score is to develop a new clinical score including the main anamnestic, and clinical features for the easy identification of pediatric FA in primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged between 0-14 years with suggestive history of food allergy

Exclusion Criteria:

* Exclusion criteria: age >14 years
* chronic systemic diseases,
* malignancy,
* immunodeficiency,
* infectious diseases,
* autoimmune diseases,
* inflammatory bowel diseases,
* celiac disease,
* metabolic and genetic diseases,
* cystic fibrosis,
* chronic pulmonary diseases,
* gastrointestinal, respiratory, urinary tract and/or cardiovascular malformations,
* neurologic and/or neuropsychiatric disorders,
* gastrointestinal tract eosinophilic disorders,
* use of immunomodulating drugs in the previous 4 months
* use of steroids and antihistamines in the previous 2 weeks

Ages: 1 Week to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects consecutively observed at the Pediatric Allergy Program, at the Department of Translational Medical Science of the University of Naples Federico II, both sex, aged 0-14 years with suggestive history of food allergy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Development of a new clinical score for the identification of pediatric FA in primary care setting | at the enrollment
  The score will include the main anamnestic and clinical features

SECONDARY OUTCOMES:
Development of a new clinical score for the identification of pediatric FA in secondary and tertiary care setting | at the enrollment
  The score will include the main anamnestic and clinical features
Validation of the new clinical NAPFA score for the identification of pediatric FA | at the enrollment
  Validation of the score on pediatric subject with suspected FA

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, MD, Principal Investigator — Department of Translational Medical Science, University of Naples Federico II
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided